CLINICAL TRIAL: NCT00823719
Title: A Single Arm, Safety and Efficacy Study of Ofatumumab in Combination With ICE or DHAP Chemotherapy in Relapsed or Refractory Aggressive Lymphoma Prior to Autologous Stem Cell Transplantation
Brief Title: Phase II Study of Ofatumumab Plus Ifosfamide, Carboplatin, Etoposide (ICE) or Dexamethasone, Cytarabine, Cisplatin (DHAP) Chemotherapy Regimen in Relapsed/ Refractory Diffuse Large B Cell Lymphoma (DLBCL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110927
Record Dates: First submitted 2009-01-08; First posted 2009-01-16 (Estimated); Results first posted 2012-09-05 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-02

CONDITIONS: Lymphoma, Large-Cell, Diffuse
Keywords: Salvage chemotherapy; relapsed; grade 3B follicular lymphoma; efficacy; safety; DHAP; ofatumumab; refractory; Non-Hodgkin's Lymphoma; Diffuse Large B Cell Lymphoma (DLBCL); Oncology; ICE; Transformed follicular lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence; Lymphoma, Non-Hodgkin; Neoplasms | interventions — ofatumumab; Ice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ofatumumab + DHAP or ICE chemotherapy regimen (Experimental): This study is a single arm study, but the Investigators are required to prospectively choose to treat all of their subjects with either ICE or DHAP chemotherapy regimens in combination with ofatumumab. Regardless of whether the subject receives ICE or DHAP chemotherapy, all subjects will receive the same ofatumumab regimen and dose.
  Interventions: Drug: ofatumumab + ICE; Drug: ofatumumab + DHAP

INTERVENTIONS:
Drug: ofatumumab + ICE — 3 cycles of treatment will be administered. Each cycle will last 21 days. ofatumumab dose: cycle 1, day 1 - 1000 milligrams (mg); cycle 1, day 8 - 1000 mg; cycle 2, day 1 and cycle 3, day 1 - 1000 mg
  ICE regimen:
  ifosfamide + mesna - 5 grams (g)/meters squared (m^2)/24 hours (hrs) continuous on day 2 of dosing cycle; carboplatin - AUC 5 (800 mg maximum) on day 2 of dosing cycle; etoposide - 100 mg/m^2 on days 1, 2 and 3 of dosing cycle.
Drug: ofatumumab + DHAP — 3 cycles of treatment will be administered. Each cycle will last 21 days. ofatumumab dose: cycle 1, day 1 - 1000 mg; cycle 1, day 8 - 1000 mg; cycle 2, day 1 and cycle 3, day 1 - 1000 mg.
  DHAP regimen:
  dexamethasone - 40 mg on days 1, 2, 3, and 4 of dosing cycle; cisplatin - 100 mg/m^2/24 hrs continuous on day 1 of dosing cycle; cytarabine - 2 g/m^2 q12 hrs (2 doses) on day 2 of dosing cycle.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ofatumumab used in combination with ifosfamide, carboplatin, etoposide (ICE) or dexamethasone, cytarabine, cisplatin (DHAP) salvage chemotherapy regimens in subjects with relapsed or refractory diffuse large B cell lymphoma (DLBCL) who are eligible for autologous stem cell transplant.

DETAILED DESCRIPTION:
Rituximab combined with anthracycline based chemotherapy is the most common first-line treatment for subjects with diffuse large B cell lymphoma (DLBCL). Subjects requiring second-line therapy will most often receive rituximab in combination with salvage chemotherapy as an induction therapy prior to autologous stem cell transplant. With rituximab being in first-line therapy, the response rates for subjects receiving rituximab plus salvage chemotherapy has significantly decreased. Treatment with ofatumumab may be able to overcome the resistance to rituximab in the second-line setting and offer improved response rates. The objective of this study is to evaluate the overall response rate of ofatumumab in combination with ICE or DHAP chemotherapy prior to autologous stem cell transplant. Additional objectives are to evaluate the complete response rate, ability to mobilize cluster of differentiation (CD)34+ cells, progression-free survival (PFS) and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with CD20 positive aggressive non-Hodgkin's lymphoma (NHL) including DLBCL, transformed follicular lymphoma (FL) & grade 3b FL.

Refractory to, or relapsed following, first-line treatment with rituximab combined with anthracycline- or anthracenedione-based chemotherapy as defined by the protocol.

* Computed tomography (CT) with involvement of 2 or more clearly demarcated lesions with a long axis > 1.5 centimeters (cm) and short axis ≥ 1.0 cm or 1 clearly demarcated lesion with a long axis >2.0 cm and short axis ≥1.0 cm.
* Baseline [18F] fluorodeoxyglucose (FDG)-positron emission tomography (PET) scans must demonstrate positive lesions compatible with CT defined anatomical tumor sites.
* Age 18 yrs or older.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
* Eligible for high dose chemotherapy and autologous stem cell transplant (ASCT).
* Resolution of toxicities from first-line therapy to a grade that in the opinion of the investigator does not contraindicate study participation.
* Signed written informed consent.

Exclusion Criteria:

* Previous cancer therapy for lymphoma, with the exception of required rituximab/ anthracycline- or anthracenedione-based chemotherapy, monotherapy rituximab prior to first-line therapy and / or as a maintenance therapy, or limited field radiotherapy (as defined by the protocol).
* Any anti-cancer therapy, except limited field radiotherapy, within 2 weeks prior to start of study therapy.
* Chronic Glucocorticoid use (limited acute use is allowed and defined by the protocol).
* History of significant cerebrovascular disease.
* Abnormal/ inadequate white blood cell (WBC) count, liver, and kidney function.
* Clinically significant cardiac disease, active or chronic infections, serious significant diseases, other cancer within last 5 years.
* Known or suspected hypersensitivity to study treatments.
* Prior treatment with anti-CD20 monoclonal antibodies, at any time, or treated with other monoclonal antibodies within 3 months prior to start of study therapy, with the exception of rituximab in both instances.
* Inability to comply with the protocol activities.
* Pregnant or lactating women or female patients of child-bearing potential (or male patients with such partners) not willing to use adequate contraception during and up to 1 year following dosing completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2009-05; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Matasar MJ, Czuczman MS, Rodriguez MA, Fennessy M, Shea TC, Spitzer G, Lossos IS, Kharfan-Dabaja MA, Joyce R, Fayad L, Henkel K, Liao Q, Edvardsen K, Jewell RC, Fecteau D, Singh RP, Lisby S, Moskowitz CH. Ofatumumab in combination with ICE or DHAP chemotherapy in relapsed or refractory intermediate grade B-cell lymphoma. Blood. 2013 Jul 25;122(4):499-506. doi: 10.1182/blood-2012-12-472027. Epub 2013 May 21. PMID 23692856

RESULTS

PARTICIPANT FLOW:
Groups:
- Ofatumumab + DHAP: Participants received 3 cycles (21 days per each cycle) of ofatumumab combined with salvage chemotherapy. Ofatumumab (1000 milligrams [mg]) was intravenously (IV) infused on Day 1 (or up to 3 days prior to Day 1) and Day 8 (+/-2 days) of Cycle 1 of the salvage chemotherapy, and then on Day 1 only of Cycles 2 and 3. The DHAP (dexamethasone, cytarabine, cisplatin) regimen (salvage chemotherapy) contained: dexamethasone (40 mg/day) administered orally or IV on Days 1, 2, 3, or 4 of each cycle; cisplatin (100 mg/square meter [m^2]/day) as an IV continuous infusion on Day 1 of each cycle; and cytarabine 2 gram (g)/m^2 over 3 hours (hr) every 12 hr (2 doses) for each infusion on Day 2 of each cycle.
- Ofatumumab + ICE: Participants received 3 cycles (21 days per each cycle) of ofatumumab combined with salvage chemotherapy. Ofatumumab (1000 mg) was IV infused on Day 1 (or up to 3 days prior to Day 1) and Day 8 (+/-2 days) of Cycle 1 of the salvage chemotherapy, and then on Day 1 only of Cycles 2 and 3. The ICE (ifosfamide, carboplatin, etoposide) regimen (salvage chemotherapy) contained: etoposide (100 mg/m^2/day) administered IV on Days 1, 2, and 3 of each cycle; carboplatin (up to 800 mg) on Day 2 of each cycle; and ifosfamide plus mesna, both at 5 g/m^2/day as an IV continuous infusion on Day 2 of each cycle.
Period: Overall Study
Arm/Group | Ofatumumab + DHAP | Ofatumumab + ICE
Started | 26 | 35
Completed | 20 | 24
Not Completed | 6 | 11
Not completed — Adverse Event | 1 | 2
Not completed — Physician Decision | 1 | 4
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Disease Progression | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ofatumumab + DHAP | Ofatumumab + ICE | Total
Number analyzed (Participants) | 26 | 35 | 61
Age Continuous [Mean (Standard Deviation); unit: Years] | 49.7 (13.79) | 53.0 (13.02) | 51.6 (13.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 15 | 20 | 35
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 2 | 2 | 4
  Asian-Central/South Asian Heritage | 1 | 0 | 1
  Asian-Japanese/East or South East Asian Heritage | 1 | 0 | 1
  White | 22 | 33 | 55
Number of participants with the indicated number of risk factors [Number; unit: participants] — The secondary age adjusted international prognostic index (SaaIPI) is assessed according to the absence or presence of 3 risk factors (RFs) at the start of Screening: Eastern Cooperative Oncology Group performance status greater than 1, lactate dehydrogenase level greater than the upper level of normal, and Ann Arbor stage II or IV disease. The presence of 0, 1, and 2/ 3 RFs corresponds to an SaaIPI score reflecting low, intermediate, and high risk of disease.
  participants
    0 or 1 | 13 | 19 | 32
    2 or 3 | 13 | 16 | 29
Number of participants in the indicated categories per best response to first line treatment [Number; unit: participants] — Late relapsers are those participants with a complete response (CR) >12 months after adequate R-CHOP-like first-line treatment. Early relapsers are those participants with a CR <= 12 months and >=28 days prior to study treatment after adequate first-line treatment. Refractory participants are those with a CR <28 days, partial response, stable disease, or progressive disease following first-line treatment.
  participants
    Late relapsers | 4 | 8 | 12
    Early relapsers/Refractory | 22 | 27 | 49

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response (OR), as Assessed by the Investigator
Description: Responders with OR included participants with complete response (CR) and partial response (PR). This was based on adequate responses from the investigator assessment after the completion of treatment. CR: complete disappearance of all detectable clinical evidence of disease and disease-related symptoms. PR: at least a 50% decrease from baseline in the sum of the product of the diameters of target lesions.
Time Frame: From Day 14 (Study Day 56) to Day 21 (approximately Study Day 63) of treatment Cycle 3, or earlier in the case of early withdrawal or missing response assessment for Cycle 3
Population: Per protocol (PP) Population: all participants who received at least one dose of ofatumumab. Participants with major protocol deviations that could have impacted the efficacy outcome, and participants not exposed to ofatumumab or without CD20+ aggressive lymphoma were excluded from assessment. CD, cluster of differentiation.
Measure: Number; unit: participants
Groups:
- Total Ofatumumab + Chemotherapy: Participants received 3 cycles (21 days per each cycle) of ofatumumab combined with salvage chemotherapy (either DHAP or ICE). Ofatumumab (1000 mg) was IV infused on Day 1 (or up to 3 days prior to Day 1) and Day 8 (+/-2 days) of Cycle 1 of the salvage chemotherapy, and then on Day 1 only of Cycles 2 and 3. DHAP contained: dexamethasone (40 mg/day) administered orally or IV on Days 1, 2, 3, or 4 of each cycle; cisplatin (100 mg/m^2/day) as an IV continuous infusion on Day 1 of each cycle; and cytarabine 2 g/m^2 over 3 hr every 12 hr (2 doses) for each infusion on Day 2 of each cycle. ICE contained: etoposide (100 mg/m^2/day) administered IV on Days 1, 2, and 3 of each cycle; carboplatin (up to 800 mg) on Day 2 of each cycle; and ifosfamide plus mesna, both at 5 g/m^2/day as an IV continuous infusion on Day 2 of each cycle.
Arm/Group | Ofatumumab + DHAP | Ofatumumab + ICE | Total Ofatumumab + Chemotherapy
Number analyzed (Participants) | 26 | 33 | 59
participants | 18 | 18 | 36
Statistical Analysis 1: Comparison: Ofatumumab + DHAP; Test type: Superiority or Other; percentage of participants = 69, 95% CI 2-sided [48.2 to 85.7] — The estimated value represents the percentage of participants with OR for participants receiving Ofatumumab + DHAP treatment
Statistical Analysis 2: Comparison: Ofatumumab + ICE; Test type: Superiority or Other; percentage of participants = 55, 95% CI 2-sided [36.4 to 71.9] — The estimated value represents the percentage of participants with OR for participants receiving Ofatumumab + ICE treatment
Statistical Analysis 3: Comparison: Total Ofatumumab + Chemotherapy; Test type: Superiority or Other; percentage of participants = 61, 95% CI 2-sided [47.4 to 73.5] — The estimated value represents the percentage of participants with OR for participants receiving Total Ofatumumab + Chemotherapy treatment

2. Secondary Outcome: Number of Participants With CR, as Assessed by the Investigator
Description: CR is defined as the complete disappearance of all detectable clinical evidence of disease and disease-related symptoms.
Time Frame: as for outcome 1
Population: PP Population
Measure: Number; unit: participants
Arm/Group | Ofatumumab + DHAP | Ofatumumab + ICE | Total Ofatumumab + Chemotherapy
Number analyzed (Participants) | 26 | 33 | 59
participants | 11 | 11 | 22

3. Secondary Outcome: Number of Participants With the Ability to Mobilize at Least 2 Million Cluster of Differentiation (CD)34+ Cells Per Kilogram (kg) From Peripheral Blood
Description: CD34+ cells are a mixture of stem cells and white blood cells of various degrees of maturity. Stem cell mobilization is the process of stimulating the hematopoietic stem cells (CD34+) to move out of the bone marrow and into the bloodstream, where they can be collected via a process called apheresis. Successful mobilization was defined as the collection of >2x10^6 CD34+ cells/kg. Only those participants, who commenced mobilization, following the administration of ofatumumab in combination with either ICE or DHAP combination chemotherapy, were assessed.
Time Frame: During treatment Cycle 2 (Study Days 22-42) and/or Cycle 3 (Study Days 43-63)
Population: Stem Cell Mobilization Population. All participants in the PP Population in whom stem cell mobilization was attempted and CD34+ cell data are available.
Measure: Number; unit: participants
Arm/Group | Ofatumumab + DHAP | Ofatumumab + ICE | Total Ofatumumab + Chemotherapy
Number analyzed (Participants) | 23 | 22 | 45
participants | 23 | 20 | 43

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the interval of time between the date of treatment start and the earlier of the date of disease progression and the date of death due to any cause. Disease progression was based on the assessments locally by investigators for the disease under study. Disease progression was based on imaging data or clinical assessment data (if radiologic assessment data were not possible or assessment was not performed).
Time Frame: as for outcome 1
Population: PP Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ofatumumab + DHAP | Ofatumumab + ICE | Total Ofatumumab + Chemotherapy
Number analyzed (Participants) | 26 | 33 | 59
days | 301.0 [152.0 to NA] — Medan survival follow-up was 208 days (6.8 months); therefore, there was not sufficient follow-up to provide an estimable upper limit of the confidence interval. | 288.0 [177.0 to NA] — Medan survival follow-up was 208 days (6.8 months); therefore, there was not sufficient follow-up to provide an estimable upper limit of the confidence interval. | 288.0 [184.0 to 349.0]

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the interval of time between the date of treatment start and the date of death due to any cause. For participants who did not die, time of death was censored at the date of last contact.
Time Frame: as for outcome 1
Population: PP Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ofatumumab + DHAP | Ofatumumab + ICE | Total Ofatumumab + Chemotherapy
Number analyzed (Participants) | 26 | 33 | 59
days | 433.0 [166.0 to NA] — Medan survival follow-up was 208 days (6.8 months); therefore, there was not sufficient follow-up to provide an estimable upper limit (UL) of the confidence interval (CI). | NA [320.0 to NA] — Half of the participants assessed did not die by the time of assessment; therefore, the median was not reached. Medan survival follow-up was 208 days (6.8 months); therefore, there was not sufficient follow-up to provide an estimable UL of the CL. | 508.0 [369.0 to NA] — Medan survival follow-up was 208 days (6.8 months); therefore, there was not sufficient follow-up to provide an estimable upper limit of the confidence interval.

6. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity, AUC(0-inf), of Ofatumumab at the First Infusion (Cycle 1, Day 1) and the Last Infusion (Cycle 3)
Description: AUC is defined as the area under the ofatumumab (Ofa) concentration-time curve as a measure of drug exposure. AUC(0-inf) is AUC from the start of infusion extrapolated to infinite time. Results are reported by first dose group and combined, as appropriate.
Time Frame: Cycle 1 Day 1 (Study Day 1; up to 1 week) and Cycle 3 (Study Day 43; up to 6 weeks)
Population: Pharmacokinetic Population: all participants (par.) exposed to ofatumumab from whom a pharmacokinetic sample was obtained and analyzed. Data for par. who switched chemotherapy regimen are not included in the summaries by chemotherapy after the switch but are included in the total summaries. Data are provided for the par. attending each visit.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*hr/mL
Arm/Group | Ofatumumab + DHAP | Ofatumumab + ICE | Total Ofatumumab + Chemotherapy
Number analyzed (Participants) | 26 | 35 | 61
µg*hr/mL
  Cycle 1 Day 1, 300 mg; n=4, 17, 21 | 34056 (0.14) | 33606 (0.15) | 33691 (0.14)
  Cycle 1 Day 1, 1000 mg; n=22, 18, 40 | 115741 (0.16) | 105898 (0.14) | 111203 (0.16)
  Cycle 3, 300 mg; n=4, 6, 10 | 222713 (0.23) | 206389 (0.06) | 212770 (0.14)
  Cycle 3, 1000 mg; n=14, 13, 30 | 258487 (0.21) | 216885 (0.17) | 232310 (0.21)
  Cycle 3, both doses; n=18, 19, 40 | 250070 (0.22) | 213514 (0.14) | 227263 (0.20)

7. Secondary Outcome: Area Under the Concentration-time Curve During the Dosing Interval (AUC(0-tau)) of Ofatumumab at the Last Infusion (Cycle 3)
Description: AUC(0-tau) is the area under the plasma concentration-time curve from time zero (0) over the dosing interval, tau, and is a measure of drug exposure. Tau is 21 days (504 hours) in this study.
Time Frame: Cycle 3 (Study Day 43; 3 weeks)
Population: Pharmacokinetic Population. Data for participants who switched chemotherapy regimen are not included in the summaries by chemotherapy after the switch but are included in the total summaries. Data are provided for the number of participants attending each visit. Results are reported by first dose group and combined, as appropriate.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*hr/mL
Arm/Group | Ofatumumab + DHAP | Ofatumumab + ICE | Total Ofatumumab + Chemotherapy
Number analyzed (Participants) | 26 | 35 | 61
µg*hr/mL
  Cycle 3, 300 mg; n=4, 6, 10 | 95112 (0.09) | 83385 (0.33) | 87891 (0.26)
  Cycle 3, 1000 mg; n=14, 13, 30 | 112676 (0.22) | 95341 (0.15) | 101948 (0.21)
  Cycle 3 both doses; n=18, 19, 40 | 108511 (0.21) | 91391 (0.22) | 98236 (0.23)

8. Secondary Outcome: Clearance (CL) of Ofatumumab
Description: CL is the clearance of drug from plasma, which is defined as the volume of plasma from which drug is removed per unit time.
Time Frame: Study Day 1 up to Study Day 85 (up to 12 weeks)
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr
Arm/Group | Ofatumumab + DHAP | Ofatumumab + ICE | Total Ofatumumab + Chemotherapy
Number analyzed (Participants) | 26 | 35 | 61
mL/hr | 8.7 (0.15) | 9.2 (0.14) | 9.0 (0.15)

9. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Ofatumumab at the First Infusion (Cycle 1 Day 1), Second Infusion (Cycle 1 Day 8), and Last Infusion (Cycle 3)
Description: Cmax is defined as the maximum concentration of drug in plasma samples for the dosing occasion.
Time Frame: Cycle 1 Day 1 (Study Day 1; up to 48 hours), Cycle 1 Day 8 (Study Day 8; up to 24 hours), Cycle 3 (Study Day 43; up to 48 hours)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Ofatumumab + DHAP | Ofatumumab + ICE | Total Ofatumumab + Chemotherapy
Number analyzed (Participants) | 26 | 35 | 61
µg/mL
  Cycle 1 Day 1, 300 mg; n=4, 17, 21 | 89.8 (0.08) | 80.0 (0.63) | 81.8 (0.56)
  Cycle 1 Day 1, 1000 mg; n=22, 18, 40 | 323 (0.40) | 268 (0.30) | 297 (0.37)
  Cycle 1 Day 8, 300 mg; n=4, 13, 17 | 245 (0.10) | 273 (0.28) | 266 (0.25)
  Cycle 1 Day 8, 1000 mg; n=21, 18, 39 | 431 (0.23) | 368 (0.21) | 401 (0.23)
  Cycle 3, 300 mg; n=4, 11, 15 | 416 (0.24) | 417 (0.26) | 417 (0.24)
  Cycle 3, 1000 mg; n=14, 14, 33 | 466 (0.31) | 397 (0.18) | 421 (0.25)
  Cycle 3, both doses; n=18, 25, 48 | 455 (0.29) | 406 (0.21) | 420 (0.25)

10. Secondary Outcome: Trough Plasma Concentration (Ctrough) of Ofatumumab Prior to Second Infusion (Cycle 1 Day 8), Third Infusion (Cycle 2), and Last Infusion (Cycle 3)
Description: Ctrough is defined as the trough plasma concentration, which is the measured concentration at the end of a dosing interval (taken directly before the start of the next infusion).
Time Frame: Cycle 1 Day 8 (Study Day 8; up to 8 hours prior to infusion start), Cycle 2 (Study Day 22; up to 7 hours prior to infusion start), Cycle 3 (Study Day 43; up to 6 hours prior to infusion start)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Ofatumumab + DHAP | Ofatumumab + ICE | Total Ofatumumab + Chemotherapy
Number analyzed (Participants) | 26 | 35 | 61
µg/mL
  Cycle 1 Day 8, 300 mg; n=4, 15, 19 | 31.8 (0.19) | 28.3 (0.93) | 29.1 (0.79)
  Cycle 1 Day 8, 1000 mg; n=19, 18, 37 | 95.8 (1.63) | 106 (0.23) | 101 (0.98)
  Cycle 2, 300 mg; n=4, 16, 20 | 112 (0.28) | 71.5 (0.81) | 78.2 (0.75)
  Cycle 2, 1000 mg; n=21, 18, 39 | 138 (0.49) | 147 (0.21) | 142 (0.38)
  Cycle 3, 300 mg; n=4, 13, 17 | 120 (0.26) | 76.7 (0.65) | 85.2 (0.60)
  Cycle 3, 1000 mg; n=18, 18, 40 | 153 (0.43) | 122 (0.45) | 134 (0.44)
  Cycle 3, both doses; n=22, 31, 57 | 146 (0.41) | 100 (0.59) | 117 (0.54)

11. Secondary Outcome: Terminal Phase Half-life (t1/2) of Ofatumumab
Description: t1/2 is defined as terminal phase half-life, which is the time required for the amount of the drug in the body to decrease by half.
Time Frame: Study Day 1 up to Study Day 85 (up to 12 weeks)
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Ofatumumab + DHAP | Ofatumumab + ICE | Total Ofatumumab + Chemotherapy
Number analyzed (Participants) | 26 | 35 | 61
hr | 595 (0.35) | 646 (0.47) | 624 (0.42)

12. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Ofatumumab
Description: Vss is the apparent volume of distribution when plasma concentrations are measured under steady state conditions. At steady state, the plasma concentration-time profile of the drug is similar after each dose.
Time Frame: Study Day 1 up to Study Day 85 (up to 12 weeks)
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Ofatumumab + DHAP | Ofatumumab + ICE | Total Ofatumumab + Chemotherapy
Number analyzed (Participants) | 26 | 35 | 61
Liters | 7.12 (0.38) | 8.13 (0.50) | 7.68 (0.46)

13. Secondary Outcome: Number of Participants Who Were Positive and Negative for Human Anti-human Antibodies (HAHA) at the Indicated Time Points
Description: Human anti-human antibodies (HAHA) indicate immune response to the administered human monoclonal antibody in a two-step assay. A positive screening result is confirmed in a second step. Negative Conclusive is subset of Negative and is a negative HAHA test result with an ofatumumab concentration <200 µg/mL in a pharmacokinetic sample collected at the same time as the HAHA sample. Data are presented when a HAHA sample was collected. WD, withdrawal; FU, follow up.
Time Frame: Study Day 1 up to approximately Study Day 63
Population: Safety Population. Data are presented for those participants who contributed a sample.
Measure: Number; unit: participants
Arm/Group | Ofatumumab + DHAP | Ofatumumab + ICE | Total Ofatumumab + Chemotherapy
Number analyzed (Participants) | 26 | 35 | 61
participants
  Positive at Day 1; n=26, 35, 61 | 0 | 0 | 0
  Negative at Day 1; n=26, 35, 61 | 26 | 35 | 61
  Positive at Early WD or FU; n=24, 30, 54 | 0 | 0 | 0
  Negative at Early WD or FU; n=24, 30, 54 | 24 | 30 | 54
  Negative conclusive at Early WD or FU; n=24, 30, 5 | 18 | 28 | 46

14. Secondary Outcome: Number of Participants With the Indicated Adverse Events (AEs) Associated With Neutropenia
Description: Neutropenia is defined as an abnormal decrease in the number of neutrophils (type of white blood cell in blood) in the blood. Febrile neutropenia is the development of fever in participants with neutropenia. Pancytopenia is defined as inadequate blood-cell formation by bone marrow, resulting in a lack of all blood-cell types.
Time Frame: Study Day 1 to approximately Study Day 63
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Ofatumumab + DHAP | Ofatumumab + ICE | Total Ofatumumab + Chemotherapy
Number analyzed (Participants) | 26 | 35 | 61
participants
  Any Event of Decreased Neutrophils; n=26, 35, 61 | 12 | 11 | 23
  Neutropenia; n=12, 11, 23 | 7 | 11 | 18
  Febrile Neutropenia; n=12, 11, 23 | 8 | 1 | 9
  Pancytopenia; n=12, 11, 23 | 1 | 0 | 1

15. Secondary Outcome: Number of Participants With the Indicated AEs Associated With Decreased Hemoglobin Counts
Description: Anaemia is defined as a pathological deficiency in the oxygen-carrying component of the blood, measured in unit volume concentrations of hemoglobin, red blood-cell volume, or red blood-cell number. Pancytopenia is defined as inadequate blood-cell formation by bone marrow, resulting in a lack of all blood-cell types.
Time Frame: Study Day 1 to approximately Study Day 63
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Ofatumumab + DHAP | Ofatumumab + ICE | Total Ofatumumab + Chemotherapy
Number analyzed (Participants) | 26 | 35 | 61
participants
  Any Event of Decreased Hemoglobin; n=26, 35, 61 | 16 | 18 | 34
  Anaemia; n=16, 18, 34 | 14 | 16 | 30
  Haemoglobin Decreased; n=16, 18, 34 | 3 | 2 | 5
  Pancytopenia; n=16, 18, 34 | 1 | 0 | 1

16. Secondary Outcome: Number of Participants With the Indicated AEs Associated With Decreased Platelet Counts
Description: Thrombocytopenia is defined as an abnormal decrease in the number of platelets in circulatory blood. Pancytopenia is defined as inadequate blood-cell formation by bone marrow, resulting in a lack of all blood-cell types.
Time Frame: Study Day 1 to approximately Study Day 63
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Ofatumumab + DHAP | Ofatumumab + ICE | Total Ofatumumab + Chemotherapy
Number analyzed (Participants) | 26 | 35 | 61
participants
  Any Event of Decreased Platelets; n=26, 35, 61 | 21 | 19 | 40
  Thrombocytopenia; n=21, 19, 40 | 20 | 19 | 39
  Pancytopenia; n=21, 19, 40 | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from Study Day 1 to approximately Study Day 63.
Arm/Group | Ofatumumab + DHAP | Ofatumumab + ICE | Total Ofatumumab + Chemotherapy
Serious Adverse Events (participants affected / at risk) | 17/26 | 7/35 | 24/61
Other Adverse Events (participants affected / at risk) | 26/26 | 35/35 | 61/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab + DHAP (N=26) | Ofatumumab + ICE (N=35) | Total Ofatumumab + Chemotherapy (N=61)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 1 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 2 | 9
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 3
Cellulitis (Infections and infestations) | 2 | 0 | 2
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 1
Device related sepsis (Infections and infestations) | 1 | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 3 | 0 | 3
Blood creatinine increased (Investigations) | 2 | 0 | 2
Blood creatinine (Investigations) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2
Caecitis (Gastrointestinal disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 1 | 3
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0 | 1
Dyskinesia (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 1 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 1
Hypersensitivity (Immune system disorders) | 2 | 0 | 2
Mental status changes (Psychiatric disorders) | 0 | 2 | 2
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab + DHAP (N=26) | Ofatumumab + ICE (N=35) | Total Ofatumumab + Chemotherapy (N=61)
Nausea (Gastrointestinal disorders) | 22 | 25 | 47
Vomiting (Gastrointestinal disorders) | 9 | 15 | 24
Constipation (Gastrointestinal disorders) | 9 | 11 | 20
Diarrhoea (Gastrointestinal disorders) | 8 | 12 | 20
Abdominal distension (Gastrointestinal disorders) | 4 | 2 | 6
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 4
Flatulence (Gastrointestinal disorders) | 3 | 0 | 3
Oral pain (Gastrointestinal disorders) | 0 | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 2
Gastritis (Gastrointestinal disorders) | 0 | 2 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 2
Toothache (Gastrointestinal disorders) | 1 | 1 | 2
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 1
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 1
Lip dry (Gastrointestinal disorders) | 0 | 1 | 1
Fatigue (General disorders) | 20 | 18 | 38
Oedema peripheral (General disorders) | 2 | 8 | 10
Oedema (General disorders) | 4 | 1 | 5
Pain (General disorders) | 5 | 0 | 5
Chest pain (General disorders) | 3 | 1 | 4
Asthenia (General disorders) | 3 | 0 | 3
Chest discomfort (General disorders) | 2 | 1 | 3
Pyrexia (General disorders) | 2 | 1 | 3
Chills (General disorders) | 1 | 1 | 2
Discomfort (General disorders) | 0 | 1 | 1
Feeling jittery (General disorders) | 1 | 0 | 1
Generalised oedema (General disorders) | 1 | 0 | 1
Local swelling (General disorders) | 1 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 1
Sensation of foreign body (General disorders) | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 11 | 13 | 24
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 14 | 19
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 9 | 11
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 8 | 11
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 10 | 10
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 6 | 7
Decreased appetite (Metabolism and nutrition disorders) | 1 | 5 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 4 | 5
Dehydration (Metabolism and nutrition disorders) | 4 | 0 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 1 | 3
Fluid overload (Metabolism and nutrition disorders) | 2 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Gout (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 18 | 34
Anaemia (Blood and lymphatic system disorders) | 12 | 15 | 27
Neutropenia (Blood and lymphatic system disorders) | 7 | 11 | 18
Lymphopenia (Blood and lymphatic system disorders) | 0 | 15 | 15
Leukopenia (Blood and lymphatic system disorders) | 0 | 13 | 13
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 9 | 6 | 15
Dizziness (Nervous system disorders) | 4 | 8 | 12
Hypoaesthesia (Nervous system disorders) | 3 | 6 | 9
Dysgeusia (Nervous system disorders) | 4 | 2 | 6
Paraesthesia (Nervous system disorders) | 1 | 5 | 6
Memory impairment (Nervous system disorders) | 0 | 4 | 4
Syncope (Nervous system disorders) | 2 | 1 | 3
Lethargy (Nervous system disorders) | 1 | 1 | 2
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 2
Burning sensation (Nervous system disorders) | 0 | 1 | 1
Neurotoxicity (Nervous system disorders) | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 1
Blood creatinine increased (Investigations) | 9 | 3 | 12
Aspartate aminotransferase increased (Investigations) | 0 | 9 | 9
Blood alkaline phosphatase increased (Investigations) | 0 | 9 | 9
Blood lactate dehydrogenase increased (Investigations) | 0 | 8 | 8
Alanine aminotransferase increased (Investigations) | 0 | 7 | 7
Weight increased (Investigations) | 6 | 0 | 6
Haemoglobin decreased (Investigations) | 0 | 2 | 2
Blood pressure increased (Investigations) | 1 | 0 | 1
Blood uric acid increased (Investigations) | 1 | 0 | 1
Brain natriuretic peptide increased (Investigations) | 1 | 0 | 1
Heart rate irregular (Investigations) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 10 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 8
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 5
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 9 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 10 | 3 | 13
Rash (Skin and subcutaneous tissue disorders) | 3 | 7 | 10
Pruritus (Musculoskeletal and connective tissue disorders) | 2 | 4 | 6
Blister (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin chapped (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Vision blurred (Eye disorders) | 2 | 2 | 4
Lacrimation increased (Eye disorders) | 0 | 3 | 3
Dry eye (Eye disorders) | 1 | 1 | 2
Blindness transient (Eye disorders) | 0 | 1 | 1
Eye pain (Eye disorders) | 1 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 1 | 1
Visual impairment (Eye disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 4 | 5 | 9
Anxiety (Psychiatric disorders) | 0 | 3 | 3
Confusional state (Psychiatric disorders) | 1 | 1 | 2
Depression (Psychiatric disorders) | 0 | 1 | 1
Hallucination, visual (Psychiatric disorders) | 0 | 1 | 1
Tearfulness (Psychiatric disorders) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 3
Urinary tract infection (Infections and infestations) | 1 | 2 | 3
Bacteraemia (Infections and infestations) | 0 | 1 | 1
Bartholin's abscess (Infections and infestations) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1
Candidiasis (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 1
Eye infection (Infections and infestations) | 0 | 1 | 1
Folliculitis (Infections and infestations) | 1 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1
Sepsis syndrome (Infections and infestations) | 0 | 1 | 1
Tooth abscess (Infections and infestations) | 1 | 0 | 1
Vulval abscess (Infections and infestations) | 1 | 0 | 1
Hypotension (Vascular disorders) | 1 | 2 | 3
Hot flush (Vascular disorders) | 1 | 1 | 2
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1
Flushing (Vascular disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 5 | 0 | 5
Ear pruritus (Ear and labyrinth disorders) | 0 | 1 | 1
Hypersensitivity (Immune system disorders) | 1 | 4 | 5
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 1
Renal impairment (Renal and urinary disorders) | 2 | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 3 | 3
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1
Aortic valve incompetence (Cardiac disorders) | 1 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2 | 2
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 1
Breast mass (Reproductive system and breast disorders) | 1 | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.